CLINICAL TRIAL: NCT04716387
Title: Estimating the Malaria Prevention Impact of New Nets: Observational Analyses to Evaluate the Evidence Generated During Piloted New Net Distributions in Mozambique
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Tropical Health LLP (Unknown); Ministry of Health, Mozambique (Other Government); Instituto Nacional de Saúde, Mozambique (Other Government); Tulane University (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 1482331
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-01

CONDITIONS: Malaria
Keywords: Long-lasting insecticidal net; LLIN; Insecticide treated net; ITN; Malaria; Epidemiology; Entomology; Anthropology; Durability monitoring; Cost-effectiveness
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chlorfenapyr ITN: These study districts will receive Interceptor G2 ITNs during the mass distribution campaign.
  Interventions: Other: Chlorfenapyr ITN
- Piperonyl butoxide ITN: This study district will receive piperonyl butoxide ITN during the mass distribution campaign.
  Interventions: Other: Piperonyl butoxide ITN
- Standard LLIN: These study districts will receive standard ITNs during the mass distribution campaign.
  Interventions: Other: Standard LLIN
- Pyriproxyfen ITN: This study district will receive Royal Guard ITNs during the mass distribution campaign.
  Interventions: Other: Pyriproxyfen ITN

INTERVENTIONS:
Other: Standard LLIN — Long-lasting insecticidal net containing alphacypermethrin, a pyrethroid insecticide, and manufactured by Shobikaa Impex Private Limited.
  Other Names: DuraNet® LLIN
  Groups: Standard LLIN
Other: Piperonyl butoxide ITN — Insecticide treated net containing permethrin, a pyrethroid, and piperonyl butoxide, an insecticide synergist, manufactured by Sumitomo Chemical.
  Other Names: Olyset®Plus ITN
  Groups: Piperonyl butoxide ITN
Other: Pyriproxyfen ITN — Insecticide treated net containing alpha-cypermethrin, a pyrethroid, and pyriproxyfen, an insect growth regulator, manufactured by Disease Control Technologies.
  Other Names: Royal Guard® ITN
  Groups: Pyriproxyfen ITN
Other: Chlorfenapyr ITN — Insecticide-treated nets containing two active ingredients: alpha-cypermethrin, a pyrethroid insecticide, and chlorfenapyr, a pyrrole insecticide, manufactured by BASF.
  Other Names: Interceptor® G2
  Groups: Chlorfenapyr ITN

SUMMARY:
The use of insecticide-treated bed nets (ITNs) has contributed to the substantial reduction in malaria cases and deaths. This progress is threatened by increasing resistance to commonly used insecticides in important mosquito vector populations. Newly developed, next-generation ITNs that use two insecticides, or an insecticide synergist and an insecticide, are effective at killing resistant mosquitoes, but large-scale uptake of these nets has been slow due to higher costs and lack of enough evidence to support broad policy recommendations.

This observational study will occur alongside a pilot distribution of next-generation ITNs in two regions of Mozambique. Over three years, data on the entomological and epidemiological impact of the different ITN types will be collected. Data collection will occur in six districts: two districts receiving the dual-active ingredient ITN Interceptor® G2 (BASF: alphacypermethrin + chlorfenapyr); one district that will receive the dual-active ingredient ITN Royal Guard® (Disease Control Technologies: alphacypermethrin + pyriproxyfen); one district receiving an ITN containing an insecticide plus an insecticide synergist , Olyset®Plus (Sumitomo Chemical: permethrin + piperonyl butoxide); and two districts receiving the standard pyrethroid-only ITNs DuraNet® (Shobikaa Impex Private Limited: alphacypermethrin). Data will be collected on malaria vector bionomics, disease epidemiology, and ITN use in order to help better demonstrate the public health value of next-generation ITNs and to support donors, policymakers, and National Malaria Control Programs in their ITN decision-making and planning processes.

DETAILED DESCRIPTION:
The World Health Organization's (WHO) 2018 World Malaria Report estimates that in 2017, 219 million cases of malaria occurred worldwide resulting in 435,000 deaths, 93% of which occurred in Africa (WHO 2018). While this represents a remarkable improvement in comparison with 2000, with malaria deaths having fallen by 40% in Africa, the downward trends in incidence and mortality stalled between 2015 and 2017. This recent failure to maintain the hard-won progress, let alone accelerate progress towards elimination, over the past three years has caused WHO to describe the global fight against malaria as being at a crossroads, calling for increased funding and highlighting the need to develop, optimize, and implement new tools to combat malaria.

Universal coverage of populations at risk with malaria vector control interventions, primarily insecticide treated nets (ITNs) and indoor residual spraying (IRS), in malaria-endemic countries is a global and national priority because of its fundamental importance for malaria control and elimination. Unfortunately, the effectiveness of these tools is threatened by the emergence and spread of pyrethroid resistance in key mosquito populations, which is now reported in more than 85% of all malaria endemic countries and poses significant risk to the future impact of these tools. Emerging evidence suggests, however, that increasing mosquito mortality and thereby continuing to reduce malaria transmission is possible in areas with pyrethroid resistance by introducing new insecticide formulations for IRS and ITNs. For example, Protopopoff et al. showed in Tanzania that the distribution of LLINs with piperonyl butoxide (PBO) plus pyrethroid reduced malaria prevalence by 13% compared to standard pyrethroid-only LLIN distribution (42% vs. 29%; p=0.0011), and Tiono et al., working in Burkina Faso, showed that the distribution of a dual active-ingredient ITN reduced clinical malaria incidence by 22% (Incidence Rate Ratio = 0.88; p=0.04) and potentially infective mosquito bites by 51% (entomological inoculation rate ratio = 0.49; p<0.0001) compared to the distribution of a standard pyrethroid-only LLIN.

While there is evidence that standard LLINs can continue to provide effective personal protection to regular net users in regions with resistant vector populations, new classes of ITNs developed to perform against pyrethroid-resistant mosquitoes have been developed, with early trials and modelling suggesting that they may provide superior protective efficacy against malaria in areas with pyrethroid-resistant vectors. Access to these new resistance-breaking ITNs is restricted by need for efficacy data for continuing policy recommendations, high prices, lack of evidence of cost effectiveness compared to pyrethroid-only LLINs, and consequent poor demand in an uncertain market. Two types of next-generation ITNs, each utilizing a different mixture of active ingredients from different insecticide classes, have recently received WHO prequalification listing demonstrating that they perform to the thresholds required of pyrethroid-only ITNs and have no known specific side effects: Interceptor G2® (IG2; by BASF SE) and Royal Guard®(RG; by Disease Control Technologies, LLC). The IG2 ITN contains a mixture of a pyrethroid (alpha-cypermethrin) and a pyrrole (chlorfenapyr), while the RG ITN contains a mixture of the same pyrethroid (alpha-cypermethrin) and an insect growth regulator (pyriproxyfen). While both net types have been subsequently registered and approved for use in Mozambique based on this WHO listing, the Roll Back Malaria Vector Control Advisory Group guidance indicates that dual active ingredient ITNs will require further epidemiological evidence before policy recommendations are made for their use in preference to pyrethroid-only ITNs in certain settings.

The Global Fund and Unitaid have developed a market shaping program for next-generation ITNs with novel insecticide formulations. Evidence on the efficacy of IG2 and RG ITNs will be generated by the project through two randomized control trials taking place in Benin and Tanzania. In addition, through this program, these next-generation ITNs will be made available to countries for incorporation into their national distribution programs as pilot distributions with the aim of determining real-world effectiveness and cost-effectiveness in different contexts. In addition to the pilot distribution of IG2s taking place in Mozambique, three other countries will be piloting next-generation ITNs as part of the New Nets project: Burkina Faso, Nigeria, and Rwanda. This research will utilize these pilot distributions to understand the cost-effectiveness of the new ITNs in the chosen settings. The NMCP in Mozambique, in discussion with the Global Fund, chose to incorporate IG2, RG, and PBO ITNs into the 2020 mass distribution campaign. This study will collect information to determine the public health impact of the RG, PBO, and IG2 ITNs in Mozambique, in comparison to two sites that will receive standard pyrethroid-only ITNs. The aim of this research is to better understand the effectiveness and cost effectiveness of IG2 and RG ITNs in Mozambique and to collect data on community uptake of the ITNs.

During the upcoming pilot implementation enhanced entomological, epidemiological, and net use data will be collected in up to six study districts: two districts receiving the dual-active ingredient ITN Interceptor® G2 (BASF: alphacypermethrin + chlorfenapyr); one district that will receive the dual-active ingredient ITN Royal Guard® (Disease Control Technologies: alphacypermethrin + pyriproxyfen); one district receiving an ITN containing an insecticide plus an insecticide synergist, Olyset®Plus (Sumitomo Chemical: permethrin + piperonyl butoxide); and two districts receiving the standard pyrethroid-only ITNs DuraNet® (Shobikaa Impex Private Limited: alphacypermethrin). Data will be analyzed and results disseminated to support the NMCP, donors, policymakers, and other national and regional stakeholders in their ITN decision-making and planning processes. Each component aims specifically to:

* Epidemiological component - measure the epidemiological impact of the new IG2 ITNs, Royal Guard ITNs, PBO ITNs, and standard ITNs in real deployment scenarios through observational studies. These studies will compare trends in (1) malaria case incidence rates passively reported to the national health system (passive case detection (PCD)) and (2) malaria infection prevalence, measured through rapid diagnostic tests (RDTs), in children aged 6 months to 5 years of age from annual cross-sectional surveys during peak transmission periods.
* Entomological component - evaluate the impact of the different net types on vector populations and biting rates, compared to standard ITNs, through mosquito surveillance data that will measure trends in species-specific (1) adult vector densities (2) indoor and outdoor human landing rates (3) estimated entomological inoculation rates and (4) insecticide resistance patterns. These entomological surveillance activities are aligned with NMCP activities and are not part of the human subject research component of this study.
* Anthropological component - map patterns of ITN usage to determine transmission risk defined as the intersection between time at risk of mosquito blood feeding and human activities not under protection of an ITN, through gathering evidence on ITN uptake and usage. The collection of reliable data on such patterns, both indoors and outdoors, becomes thus an essential component of the evaluation of the ITN pilots for both modeling and contextual analysis of impact.
* Durability monitoring - monitoring of standard, IG2, RG and PBO ITNs in one district each, prospectively measuring physical durability, attrition, and chemical durability.
* Costing and cost-effectiveness component - estimate the cost and cost-effectiveness of IG2, RG and PBO ITNs in Mozambique through data on the price of the product, delivery and deployment costs, and product effectiveness based on case incidence rates measured during the epidemiological component of this study. Additionally, mean costs per case averted that might occur in other contexts will be modeled and incorporated into the cost-effectiveness evaluations.

ELIGIBILITY:
Inclusion Criteria:

* All suspected malaria cases (fevers) that self-present to the national health system and are counted in the district health surveillance systems (Passive data collection)
* Households in the district (Cross-sectional)
* Residents of the household visited (Cross-sectional
* Questionnaire: parent or guardian giving written informed consent (cross-sectional)
* Malaria screening: child aged 6 to 59 months from the above consenting household.

Exclusion Criteria:

* District non-residents
* Malaria screening: history of recent (within one month) malaria infection or treatment with anti-malarial medication (cross-sectional)
* Parents or guardians who have not yet reached age of consent (18 years) and their children will not be included in study activities requiring consent.
* Head of household unwilling and/or unable to give consent

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study districts are located in Niassa and Zambezia provinces of northern Mozambique and Manica, Sofala, and Tete provinces in western Mozambique. The study districts, Mandima, Cuamba, Gurue, Changara, Guro, and Chemba will receive enhanced data collection. In addition, routine entomological and epidemiological data from all districts in these provinces will be used to compare trends. The study districts have similar malaria transmission dynamics. Routine data provided by in-country stakeholders show that these districts are comparable in underlying malaria prevalence, incidence, vector species composition, and insecticide resistance status, as well as general climate and geographic similarities.
Sampling Method: Probability Sample
Enrollment: 8726 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Cumulative malaria incidence | August 2020 to December 2022
  Malaria incidence measured through passive case detection at health facilities in each district. This measure accounts for symptomatic cases self-reporting to the formal health system for care.

SECONDARY OUTCOMES:
Vectors species composition | August 2020 to December 2022
  All Anopheles mosquitoes sampled during human landing collections (HLC) will be identified morphologically to species group
Species-specific population densities | August 2020 to December 2022
  Based on Anopheles mosquitoes sampled during HLCs.
Biting behaviors | August 2020 to December 2022
  Based on Anopheles mosquitoes sampled during HLCs.
Estimated entomological inoculation rates | August 2020 to December 2022
  Based on Anopheles mosquitoes sampled during HLCs.
Insecticide resistance profile | August 2020 to December 2022
  Measurement of kdr and ace-1 mutation frequencies, WHO tube bioassays at minimum and CDC bottle bioassays to characterize insecticide resistance intensity
Parasite prevalence in children 6-59 months | August 2020, August 2021, August 2022
  Prevalence calculated from cross-sectional surveys conducted during the peak transmission season.
Net use characteristics | August 2020 to December 2022
  Mapping the social determinants of intervention impact and transmission risk as the intersection of time at risk of mosquito blood feeding and human activities not under the protection of an ITN by gathering data on ITN uptake through structured observations
Cost-effectiveness measures | August 2020 to December 2022
  Estimated cost and cost-effectiveness through measurements of delivery and commodity costs collected through interviews and written questionnaires of New Nets Project stakeholders and representatives of the NMCP, implementing partners, procurement agencies, and manufacturing firms, in combination with effect estimates for interventions.
Physical durability monitoring | January 2021, July 2021, June 2022
  Assess the physical durability of ITNs after two years of use.
Insecticide durability monitoring | January 2021, July 2021, June 2022
  Assess the insecticidal effectiveness of ITNs after two years of use.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wagman, PhD, Principal Investigator — PATH
Locations (1):
- Programa Nacional de Controle da Malaria, Ministry of Health, Maputo, Mozambique

REFERENCES:
- [Background] Abilio AP, Marrune P, de Deus N, Mbofana F, Muianga P, Kampango A. Bio-efficacy of new long-lasting insecticide-treated bed nets against Anopheles funestus and Anopheles gambiae from central and northern Mozambique. Malar J. 2015 Sep 17;14:352. doi: 10.1186/s12936-015-0885-y. PMID 26377825
- [Background] Alonso P, Noor AM. The global fight against malaria is at crossroads. Lancet. 2017 Dec 9;390(10112):2532-2534. doi: 10.1016/S0140-6736(17)33080-5. Epub 2017 Nov 29. No abstract available. PMID 29195688
- [Background] Bass C, Nikou D, Donnelly MJ, Williamson MS, Ranson H, Ball A, Vontas J, Field LM. Detection of knockdown resistance (kdr) mutations in Anopheles gambiae: a comparison of two new high-throughput assays with existing methods. Malar J. 2007 Aug 13;6:111. doi: 10.1186/1475-2875-6-111. PMID 17697325
- [Background] Bhatt S, Weiss DJ, Cameron E, Bisanzio D, Mappin B, Dalrymple U, Battle K, Moyes CL, Henry A, Eckhoff PA, Wenger EA, Briet O, Penny MA, Smith TA, Bennett A, Yukich J, Eisele TP, Griffin JT, Fergus CA, Lynch M, Lindgren F, Cohen JM, Murray CLJ, Smith DL, Hay SI, Cibulskis RE, Gething PW. The effect of malaria control on Plasmodium falciparum in Africa between 2000 and 2015. Nature. 2015 Oct 8;526(7572):207-211. doi: 10.1038/nature15535. Epub 2015 Sep 16. PMID 26375008
- [Background] Fornadel CM, Norris LC, Franco V, Norris DE. Unexpected anthropophily in the potential secondary malaria vectors Anopheles coustani s.l. and Anopheles squamosus in Macha, Zambia. Vector Borne Zoonotic Dis. 2011 Aug;11(8):1173-9. doi: 10.1089/vbz.2010.0082. Epub 2010 Dec 13. PMID 21142969
- [Background] Kleinschmidt I, Bradley J, Knox TB, Mnzava AP, Kafy HT, Mbogo C, Ismail BA, Bigoga JD, Adechoubou A, Raghavendra K, Cook J, Malik EM, Nkuni ZJ, Macdonald M, Bayoh N, Ochomo E, Fondjo E, Awono-Ambene HP, Etang J, Akogbeto M, Bhatt RM, Chourasia MK, Swain DK, Kinyari T, Subramaniam K, Massougbodji A, Oke-Sopoh M, Ogouyemi-Hounto A, Kouambeng C, Abdin MS, West P, Elmardi K, Cornelie S, Corbel V, Valecha N, Mathenge E, Kamau L, Lines J, Donnelly MJ. Implications of insecticide resistance for malaria vector control with long-lasting insecticidal nets: a WHO-coordinated, prospective, international, observational cohort study. Lancet Infect Dis. 2018 Jun;18(6):640-649. doi: 10.1016/S1473-3099(18)30172-5. Epub 2018 Apr 9. PMID 29650424
- [Background] Koekemoer LL, Kamau L, Hunt RH, Coetzee M. A cocktail polymerase chain reaction assay to identify members of the Anopheles funestus (Diptera: Culicidae) group. Am J Trop Med Hyg. 2002 Jun;66(6):804-11. doi: 10.4269/ajtmh.2002.66.804. PMID 12224596
- [Background] Protopopoff N, Mosha JF, Lukole E, Charlwood JD, Wright A, Mwalimu CD, Manjurano A, Mosha FW, Kisinza W, Kleinschmidt I, Rowland M. Effectiveness of a long-lasting piperonyl butoxide-treated insecticidal net and indoor residual spray interventions, separately and together, against malaria transmitted by pyrethroid-resistant mosquitoes: a cluster, randomised controlled, two-by-two factorial design trial. Lancet. 2018 Apr 21;391(10130):1577-1588. doi: 10.1016/S0140-6736(18)30427-6. Epub 2018 Apr 11. PMID 29655496
- [Background] Ranson H, N'guessan R, Lines J, Moiroux N, Nkuni Z, Corbel V. Pyrethroid resistance in African anopheline mosquitoes: what are the implications for malaria control? Trends Parasitol. 2011 Feb;27(2):91-8. doi: 10.1016/j.pt.2010.08.004. Epub 2010 Sep 16. PMID 20843745
- [Background] Scott JA, Brogdon WG, Collins FH. Identification of single specimens of the Anopheles gambiae complex by the polymerase chain reaction. Am J Trop Med Hyg. 1993 Oct;49(4):520-9. doi: 10.4269/ajtmh.1993.49.520. PMID 8214283
- [Background] Sherrard-Smith E, Griffin JT, Winskill P, Corbel V, Pennetier C, Djenontin A, Moore S, Richardson JH, Muller P, Edi C, Protopopoff N, Oxborough R, Agossa F, N'Guessan R, Rowland M, Churcher TS. Systematic review of indoor residual spray efficacy and effectiveness against Plasmodium falciparum in Africa. Nat Commun. 2018 Nov 26;9(1):4982. doi: 10.1038/s41467-018-07357-w. PMID 30478327
- [Background] Tiono AB, Ouedraogo A, Ouattara D, Bougouma EC, Coulibaly S, Diarra A, Faragher B, Guelbeogo MW, Grisales N, Ouedraogo IN, Ouedraogo ZA, Pinder M, Sanon S, Smith T, Vanobberghen F, Sagnon N, Ranson H, Lindsay SW. Efficacy of Olyset Duo, a bednet containing pyriproxyfen and permethrin, versus a permethrin-only net against clinical malaria in an area with highly pyrethroid-resistant vectors in rural Burkina Faso: a cluster-randomised controlled trial. Lancet. 2018 Aug 18;392(10147):569-580. doi: 10.1016/S0140-6736(18)31711-2. Epub 2018 Aug 10. PMID 30104047
- [Background] Weill M, Malcolm C, Chandre F, Mogensen K, Berthomieu A, Marquine M, Raymond M. The unique mutation in ace-1 giving high insecticide resistance is easily detectable in mosquito vectors. Insect Mol Biol. 2004 Feb;13(1):1-7. doi: 10.1111/j.1365-2583.2004.00452.x. PMID 14728661